CLINICAL TRIAL: NCT02611375
Title: Conditioning Neural Circuits to Improve Upper Extremity Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shepherd Center, Atlanta GA (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS-668
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Spinal Cord Injury; Tetraplegia
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- tDCS + FTP group (Experimental): This group of individuals with tetraplegia will receive transcranial direct current stimulation (tDCS) over the hand area of their primary motor cortex (M1). Stimulation at 2mA will be applied for 20 minutes while subjects complete a total of 1 hour of functional task practice (FTP) per session. (Only 20 minutes of functional task practice be be performed with stimulation on). 3 sessions will be completed per week for 4 weeks.
  Interventions: Other: transcranial direct current stimulation
- PNSS + FTP group (Active Comparator): This group of individuals with tetraplegia will receive peripheral nerve somatosensory stimulation (PNSS) to the median nerve of the primary hand being trained. Stimulation will be set to elicit a sensory - not motor - response. Stimulation will be performed concurrently with the entire functional task practice (FTP) session. 3 sessions will be completed per week for 4 weeks.
  Interventions: Other: peripheral nerve somatosensory stimulation
- sham tDCS + FTP group (Active Comparator): This group of individuals with tetraplegia will receive sham transcranial direct current stimulation (tDCS) over the hand area of their primary motor cortex (M1) alongside functional task practice. Stimulation will be briefly turned on at the beginning of FTP and again after 20 minutes of practice in order to create a sham effect and maintain blinding of the participants. 3 sessions will be completed per week for 4 weeks.
  Interventions: Other: sham transcranial direct current stimulation

INTERVENTIONS:
Other: transcranial direct current stimulation — High-definition transcranial direct current stimulation is applied over the hand area of the primary motor cortex (M1). Parameters= 2mA for 20 minutes. Functional task practice will be completed concurrently with tDCS and for approximate 40 minutes after the stimulation stops.
  Other Names: tDCS
  Arms: tDCS + FTP group
Other: peripheral nerve somatosensory stimulation — Electrical stimulation will be applied to the median nerve of the primary hand being trained at parameters that elicit a sensory but not motor response (called "peripheral nerve somatosensory stimulation"). Stimulation parameters are 100Hz with a 250uS pulse width. Stimulation intensity will vary between 1-10mA per participant. Stimulation will be applied for 1 hour and functional task practice will be completed concurrent with the stimulation.
  Arms: PNSS + FTP group
Other: sham transcranial direct current stimulation — During sham transcranial direct current stimulation (tDCS), a sham tDCS device will be used along with functional task practice. The sham tDCS unit will be used for the first 20 minutes of FTP, followed by an additional 40 minutes of FTP.
  Arms: sham tDCS + FTP group

SUMMARY:
Non-invasive brain stimulation has gained increasing popularity and research support over the past several years. Recent research indicates that it might have benefits for improving hand function in people with spinal cord injury. The purpose of this study is to evaluate the effects of a type of non-invasive brain stimulation, known as tDCS, on hand function.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is a technique in which low intensity electrical current is applied over the skull in order to excite the underlying brain tissue. It has been studied in many populations (stroke, spinal cord injury, learning disability, migraine, memory) and may be a useful counterpart to traditional rehabilitation of neurological injuries. Preliminary studies from members of the investigator's lab group have indicated beneficial, single-session effects of tDCS on hand function in people with spinal cord injury. Longer-term, multi-session trials are now warranted.

Another approach that has research support for augmenting the effects of hand function training is peripheral nerve somatosensory stimulation (PNSS). Unlike tDCS, which excites brain tissue directly, PNSS excites the brain via an indirect approach. Members of the investigators' lab have found the combination of PNSS and fine motor training to be more effective in improving hand function than either intervention alone. Multi-session trials of PNSS have been conducted; however it has not yet been compared with another clinically accessible adjunctive therapy, like tDCS, in a multi-session trial.

The investigators plan to study the comparative effects of tDCS and hand function training to PNSS and hand function training and hand function training alone in people with neck-level spinal cord injuries. People with both acute/subacute (<6 months post-injury) and chronic (>1 year post-injury) injuries will be enrolled, in order to look at responses to tDCS at different stages of recovery.

Before beginning training, participants will complete approximately three hours of testing of their arm/hand function and self-reported perception of their overall function. Participants will then be randomly assigned to receive either tDCS, PNSS, or sham tDCS in combination with personalized fine motor training. This training will take place 3 times/week, for a total of 3 hours of training/week, for 4 weeks. Fine motor training will be based on principles that have been shown to optimize neuroplasticity (changes in the brain and/or spinal cord), yet customized, in order to allow participants to work towards individualized goals. At the end of 4 weeks, participants will complete a three-hour post-test using the same measures as before to examine any changes in arm and hand function. Participants will be asked to return to Shepherd Center 4 - 6 weeks following the post-intervention assessment to complete the post-intervention assessment.

ELIGIBILITY:
Inclusion Criteria:

* Be 18-65 years of age
* Have a cervical (neurological level C1-C8) SCI that occurred either <6 months ago (subacute) or >1 year (chronic) prior to the time of enrollment
* For subjects with acute/subacute SCI: the injury must be a traumatic injury (i.e. not the result of illness or a condition within the body)
* Have ISNCSCI severity classification (A, B, C or D)
* Have self-reported limitations in arm and hand function in at least one upper limb (a GRASSP quantitative score of no more than 26/30 in the hand that is the focus of treatment)
* Have the ability to pick up objects with at least one hand without using assistive devices (a GRASSP quantitative score of at least 4/30 in the hand that is the focus of treatment)
* Have shoulder strength lift an arm up to chest level
* Have the ability to sit for at least one hour at a time (e.g. good skin integrity, stable blood pressure)
* For subjects with acute/subacute SCI: adequate time remaining in their treatment at Shepherd Center to allow 5 weeks of participation
* For subjects with chronic SCI: active hand function is required (see Pre-intervention assessment) reliable transportation in order to complete the intervention in its entirety
* Ability and willingness to consent and authorize use of personal health information

Exclusion Criteria:

* Pacemaker or a metal implant in the head
* Current pregnancy
* Severe shoulder weakness, injury, or pain that contraindicates repetitive fine motor training
* Lower motor neuron damage (as documented in medical record, per participant report, or as noted by in-person screening)
* Severe hypersensitivity or pain of the arm/hand
* Severe contractures of the arm/hand that would limit participation in fine motor training
* Prior tendon or nerve transfer surgery
* Have a history of seizures
* Have a history of frequent or severe headaches

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Change in Quantitative Prehension Ability (GRASSP subtest) | Baseline, 1 week post-intervention, 4-6 weeks post-intervention
  Pre-, post-, and follow-up upper extremity impairment and function

SECONDARY OUTCOMES:
Change in Upper Extremity Strength (Grip and Pinch Strength) | Baseline, 1 week post-intervention, 4-6 weeks post-intervention
  Pre-, post-, and follow-up upper extremity impairment and function
Change in Upper Extremity Sensation (Semmes-Weinstein) | Baseline, 1 week post-intervention, 4-6 weeks post-intervention
  Pre-, post-, and follow-up upper extremity impairment and function
Change in Perceived Upper Extremity Performance & Satisfaction (COPM) | Baseline, 1 week post-intervention, 4-6 weeks post-intervention
  Pre-, post-, and follow-up self-perceived upper extremity function
Short-term change in Quantitative Prehension Ability (Abbreviated GRASSP) subtest) | weekly during 4-week treatment period
  weekly assessment of upper extremity function
Classification of Upper Extremity Function (BHUEF) | Baseline, 1 week post-intervention, 4-6 weeks post-intervention
  Pre-, post-, and follow-up upper extremity impairment and function
Detection of Hand Muscle Activation (subclinical EMG) | Baseline, 1 week post-intervention, 4-6 weeks post-intervention
  Pre-, post-, and follow-up upper extremity impairment and function
Change in Perceived Quality of Life (SCI QoL Basic Data Set) | Baseline, 1 week post-intervention, 4-6 weeks post-intervention
  Pre-, post-, and follow-up self-perceived quality of life rating
Change in Cortical Excitability (motor evoked potentials) | Baseline, 1 week post-intervention, 4-6 weeks post-intervention
  Pre-, post-, and follow-up neural excitability
Change in Spinal Reflex Excitability (joint threshold angle) | Baseline, 1 week post-intervention, 4-6 weeks post-intervention
  Pre-, post-, and follow-up neural excitability

CONTACTS AND LOCATIONS:
Overall Officials: Edelle C Field-Fote, PT, PhD, Principal Investigator — Shepherd Center, Atlanta GA
Locations (1):
- Shepherd Center, Inc., Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Gomes-Osman J, Field-Fote EC. Bihemispheric anodal corticomotor stimulation using transcranial direct current stimulation improves bimanual typing task performance. J Mot Behav. 2013;45(4):361-7. doi: 10.1080/00222895.2013.808604. Epub 2013 Jun 24. PMID 23796102
- [Background] Anderson KD. Targeting recovery: priorities of the spinal cord-injured population. J Neurotrauma. 2004 Oct;21(10):1371-83. doi: 10.1089/neu.2004.21.1371. PMID 15672628
- [Background] Biering-Sorensen F, Bryden A, Curt A, Friden J, Harvey LA, Mulcahey MJ, Popovic MR, Prochazka A, Sinnott KA, Snoek G. International spinal cord injury upper extremity basic data set. Spinal Cord. 2014 Sep;52(9):652-7. doi: 10.1038/sc.2014.87. Epub 2014 Jun 3. PMID 24891012
- [Background] Beekhuizen KS, Field-Fote EC. Massed practice versus massed practice with stimulation: effects on upper extremity function and cortical plasticity in individuals with incomplete cervical spinal cord injury. Neurorehabil Neural Repair. 2005 Mar;19(1):33-45. doi: 10.1177/1545968305274517. PMID 15673842
- [Background] Hoffman LR, Field-Fote EC. Cortical reorganization following bimanual training and somatosensory stimulation in cervical spinal cord injury: a case report. Phys Ther. 2007 Feb;87(2):208-23. doi: 10.2522/ptj.20050365. Epub 2007 Jan 9. PMID 17213410
- [Background] Hoffman LR, Field-Fote EC. Functional and corticomotor changes in individuals with tetraplegia following unimanual or bimanual massed practice training with somatosensory stimulation: a pilot study. J Neurol Phys Ther. 2010 Dec;34(4):193-201. doi: 10.1097/NPT.0b013e3181fbe692. PMID 21084920
- [Background] Gomes-Osman J, Field-Fote EC. Cortical vs. afferent stimulation as an adjunct to functional task practice training: a randomized, comparative pilot study in people with cervical spinal cord injury. Clin Rehabil. 2015 Aug;29(8):771-82. doi: 10.1177/0269215514556087. Epub 2014 Nov 7. PMID 25381344
- [Background] Birkenmeier RL, Prager EM, Lang CE. Translating animal doses of task-specific training to people with chronic stroke in 1-hour therapy sessions: a proof-of-concept study. Neurorehabil Neural Repair. 2010 Sep;24(7):620-35. doi: 10.1177/1545968310361957. Epub 2010 Apr 27. PMID 20424192
- [Background] Charlifue S, Post MW, Biering-Sorensen F, Catz A, Dijkers M, Geyh S, Horsewell J, Noonan V, Noreau L, Tate D, Sinnott KA. International Spinal Cord Injury Quality of Life Basic Data Set. Spinal Cord. 2012 Sep;50(9):672-5. doi: 10.1038/sc.2012.27. Epub 2012 Mar 27. PMID 22450884
- [Background] Kalsi-Ryan S, Beaton D, Curt A, Duff S, Popovic MR, Rudhe C, Fehlings MG, Verrier MC. The Graded Redefined Assessment of Strength Sensibility and Prehension: reliability and validity. J Neurotrauma. 2012 Mar 20;29(5):905-14. doi: 10.1089/neu.2010.1504. Epub 2011 Aug 12. PMID 21568688
- [Background] Lohse KR, Boyd LA, Hodges NJ. Engaging Environments Enhance Motor Skill Learning in a Computer Gaming Task. J Mot Behav. 2016;48(2):172-82. doi: 10.1080/00222895.2015.1068158. Epub 2015 Aug 21. PMID 26296097
- [Background] Velstra IM, Curt A, Frotzler A, Abel R, Kalsi-Ryan S, Rietman JS, Bolliger M. Changes in Strength, Sensation, and Prehension in Acute Cervical Spinal Cord Injury: European Multicenter Responsiveness Study of the GRASSP. Neurorehabil Neural Repair. 2015 Sep;29(8):755-66. doi: 10.1177/1545968314565466. Epub 2015 Jan 7. PMID 25567122